CLINICAL TRIAL: NCT07226258
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose Study to Assess the Safety and Efficacy of SL1002 Injectable for the Treatment of Knee Pain in Patients With Osteoarthritis of the Knee
Brief Title: Phase III Study to Assess the Safety and Efficacy of SL1002 for Osteoarthritis Knee Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Saol Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SL-1010-02
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis Knee Pain
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SL1002 (Experimental): SL1002
  Interventions: Drug: SL1002
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: SL1002 — SL1002 injectable solution
  Arms: SL1002
Drug: Normal Saline — Normal Saline
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Single Dose Study to Assess the Safety and Efficacy of SL1002 for the Treatment of Knee Pain in Patients with Osteoarthritis of the Knee.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of a single treatment of SL1002 compared to placebo for the treatment of knee pain associated with mild to moderate osteoarthritis.

ELIGIBILITY:
Inclusion Criteria includes:

1. Male or female patients ≥ 40 years of age
2. Body Mass Index (BMI) limits
3. Chronic knee pain resulting from osteoarthritis
4. Kellgren-Lawrence Grade 2 (mild) or Grade 3 (moderate)
5. Baseline KOOS pain
6. Patients taking baseline analgesics
7. Diagnostic nerve block response
8. Compliance with identified study requirements

Exclusion Criteria includes:

1. Non-OA inflammatory arthritis
2. Confounding elements
3. Lower limb amputation.
4. Specified alternate historic treatments
5. Identified underlying physiologic or psychosocial conditions
6. Patient Health Questionnaire
7. Moderate to severe hepatic impairment
8. Moderate to severe renal impairment
9. Identifiable baseline medications
10. Protocol compliance requirements
11. Known allergies or hypersensitivity to identified agents
12. Identified alcohol or drug abuse history
13. Identified underlying physical exam findings: ECG abnormalities or vital sign abnormalities during study screening per investigator assessment
14. Identified underlying abnormal laboratory results

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 12 in the Weekly Mean of the Average Daily Pain Intensity While Walking | Baseline to week 12
  The pain intensity score is measured using a numeric rating scale (NRS)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - DBPS Research, LLC, Greenwood Village, Colorado
  - International Spine, Pain & Performance Center, Washington D.C., District of Columbia
  - Prime Medical Research, Coral Gables, Florida
  - Conquest Research, LLC, Orlando, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Queen City Clinical Research, PLLC, Charlotte, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Pacific Sports and Spine, Eugene, Oregon
  - University Orthopedics Center, Altoona, Pennsylvania
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - HD Research, First Surgical Hospital (FSH), Bellaire, Texas
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Virginia iSpine Physicians, PC, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No